CLINICAL TRIAL: NCT03105739
Title: Timing of Withdrawal of the Laryngeal Mask Airway (LMA) in Children: Early or Late Removal?
Brief Title: Timing of Withdrawal of the Laryngeal Mask Airway (LMA) in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital d'enfants Béchir-Hamza (Other)
Responsible Party: Principal Investigator, Dr Sonia ben khalifa (PhD), Head of Anesthesia and Intensive Care Department, Hôpital d'enfants Béchir-Hamza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LMA-001
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Laryngeal Mask Airway Removal; Respiratory Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthetised (Experimental): LMA removal once the halogenated anesthetic turned off
  Interventions: Other: LMA removal
- Awake (Active Comparator): LMA removal once the patient fully regained consciousness
  Interventions: Other: LMA removal

INTERVENTIONS:
Other: LMA removal — According to randomization, LMA device was removed at the end of surgery, either in deeply anesthetised patients or after consciousness recovery.

SUMMARY:
The purpose of this prospective, randomized study was to compare the incidence of adverse events associated with removal of the LMA either in deeply anesthetised or awake patients.

DETAILED DESCRIPTION:
Written informed consent was obtained from parents for this prospective, randomized study conducted on children scheduled for minor surgery. Anesthesia was induced with sevoflurane, supplemented with propofol (3mg/kg) then maintained with nitrous oxide and sevoflurane 2-4% in oxygen. Analgesia was insured by peripheral nerve blocks. Included children were randomized into 2 groups:

* Awake: the LMA was left in place until the patient fully regained consciousness
* Deeply anesthetised: the LMA was immediately removed once the halogenated anesthetic turned off, and ventilation using facial mask was carried until spontaneous ventilation recovery.

Respiratory complications that occurred during LMA removal until 20 minutes afterwards were recorded. Children with respiratory history and those for whom peripheral nerve blocks failed, were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for minor surgery

Exclusion Criteria:

* None

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2016-10-05; Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Occurence of respiratory adverse events | from LMA removal to 20 minutes afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Ben Khalifa, PhD, Principal Investigator
Locations (1):
- Hôpital d'Enfants Béchir Hamza, Bab Saadoun, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No